CLINICAL TRIAL: NCT02121405
Title: Randomized Trial of Primary Surgery Followed Selective Radiochemotherapy Versus Conventional Preoperative Radiochemotherapy for Locally Advanced Rectal Cancer With MRI Negative Circumferential Margin
Brief Title: Randomized Trial of Primary Surgery Followed Selective Radiochemotherapy for Rectal Cancer With MRI Negative CRM
Acronym: PSSR
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB stopped this trial due to the difference of 3-year DFS's rate between two groups more than 5% at the interim analysis in July 2021.
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Ding Ke-Feng, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRCCZ-R01
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Neoplasm; Effects of Radiation Therapy; Effects of Chemotherapy; Surgery
MeSH Terms: conditions — Colorectal Neoplasms; Radiation Injuries | interventions — Radiotherapy; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primary surgery (Experimental): The patients receive primary rectectomy including anterior resection or abdominoperineal resection by open or laparoscopy with TME. To patients with pathological confirmed positive circumferential margin (CRM), postoperative concurrent radiochemotherapy is required that starts in 3 months post operation with capecitabine. Capecitabine and Oxaliplatin (CapeOx) chemotherapy starts in 4 weeks post operation to total of 6 cycles/18 weeks. To patients with pathological confirmed negative CRM, radiotherapy is omitted. The stage III patients receive 8 cycles/6 months CapeOx chemotherapy. The stage II patients with low microsatellite instability (MSI) receive 8 cycles/6 months Capecitabine chemotherapy. The stage II patients with high MSI and stage I patients do not receive adjuvant therapy.
  Interventions: Procedure: Rectectomy; Radiation: Radiotherapy; Drug: Capecitabine; Drug: Oxaliplatin
- Preoperative radiochemotherapy (Active Comparator): All of the patients receive conventional concurrent radiochemotherapy with capecitabine for 5 weeks. Then all of the patients receive 2 cycles/6 weeks capecitabine ± Oxaliplatin chemotherapy. Patients receive rectectomy including anterior resection or abdominoperineal resection by open or laparoscopy with total mesorectal excision 8 weeks post radiotherapy. All of the patients receive 5 cycles/15 weeks capecitabine ± Oxaliplatin adjuvant chemotherapy. The use of Oxaliplatin depends on the doctor's decision.
  Interventions: Procedure: Rectectomy; Radiation: Radiotherapy; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Procedure: Rectectomy — Include anterior resection or abdominoperineal resection by open or laparoscopy with Total Mesorectal Excision (TME).
Radiation: Radiotherapy — 45-50 Gy in 25-28 fractions to the pelvis. After 45 Gy a tumor bed boost with a 2 cm margin of 5.4 Gy in 3 fractions for preoperative cancers or 5.4-9.0 Gy in 3-5 fractions for postoperative cancers could be considered. Radiotherapy is used only for patients with pathological confirmed positive circumferential margin in Group primary surgery. Radiotherapy is used to all of the patients in Group preoperative radiochemotherapy.
Drug: Capecitabine — Capecitabine 825 mg/m2 twice daily 5 or 7 days/week with concurrent radiotherapy in Group primary surgery and Group preoperative radiochemotherapy. Capecitabine 1250 mg/m2 twice daily 1-14 every 3 weeks to a total of 6 weeks after preoperative radiochemotherapy in Group preoperative radiochemotherapy. Capecitabine 1250 mg/m2 twice daily 1-14 every 3 weeks to a total of 6 months postoperative therapy for a part of stage II patients in Group of primary surgery. Capecitabine 1000 mg/m2 twice daily 1-14 every 3 weeks with oxaliplatin day 1 to a total of 6 months postoperative therapy for stage III patients in Group of primary surgery.
  Other Names: Xeloda
Drug: Oxaliplatin — Oxaliplatin 130 mg/m2 over 2 hours, day 1, with capecitabine every 3 weeks. Repeat every 3 weeks to total of 6 months postoperative therapy.
  Other Names: Eloxatin

SUMMARY:
The purpose of this study is to determine whether primary radiotherapy can be omitted for the locally advanced rectal cancer with Magnetic Resonance Imaging (MRI) negative circumferential margin.

DETAILED DESCRIPTION:
The preoperative radiochemotherapy with fluorouracil followed surgery is the standard therapy for patients with locally advanced rectal cancer. However, the necessity of radiotherapy has been questioned for a long time especially for patients with enough circumferential margins. Moreover, indiscriminate radiotherapy will result Irreversible ovarian dysfunction for female. In the past decade, there were two major progresses for colorectal cancer. Firstly, oxaliplatin with fluorouracil has become the standard adjuvant chemotherapy for advanced colon cancer. Oxaliplatin improved the survival of colon cancer patients than single fluorouracil. Our experience showed that oxaliplatin with fluorouracil could improve the prognosis of rectal cancer without radiotherapy. It has been proven that oxaliplatin should not add to radiotherapy for rectal cancer. However, whether oxaliplatin can replace radiotherapy for certain rectal cancer patients is still unknown. Secondly, Magnetic Resonance Imaging (MRI) has been proven that can predict the circumferential margin status for rectal cancer. Now, preoperative MRI scan can recognize the rectal cancer patients with low recurrence risk. The radiotherapy may be omitted to the patients with low recurrence risk. This study is a randomized controlled trial to compare the 3-year disease-free survival (DFS) differences of group of experiment (the patients receive primary surgery followed selective radiochemotherapy) and group of control (the patients receive indiscriminate preoperative radiochemotherapy followed surgery) for locally advanced rectal cancer with negative MRI circumferential margin.

ELIGIBILITY:
Inclusion Criteria:

* Rectal adenocarcinoma or mucinous adenocarcinoma that is 6-12 cm from the anal verge.
* MRI scan confirmed cT3N0 or cT4aN0 or cT1-4aN+ mid rectal cancer (6-12cm from the anal verge).
* MRI scan confirmed more than 1 mm circumferential margin.
* Age 18-75 years old.
* Without distant metastasis.

Exclusion Criteria:

* Malignant history.
* Contraindications of MRI scan.
* Contraindications of radiotherapy.
* Contraindications of chemotherapy.
* Pregnancy.
* Multidisciplinary team thinks that the patient is unsuitable to take part in research (For example, there are obvious regional lymph nodes involved in low rectal cancer patients who are thought with high risk of recurrence).
* Refuse to take part in research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | Three years from the date of randomization

SECONDARY OUTCOMES:
The rate of positive circumferential resection margin | 1 day of postoperative pathological examination.
Quality of life by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C(core) 30 and QLQ-CR(colorectal) 29 forms | Baseline before any treatment,3 months post operation, 1 year post operation
Overall survival | Five years from the date of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Feng Ding, M.D., Principal Investigator — The Second Affiliated Hospital Zhejiang University Medical School
Locations (7):
- China (7):
  - Union Hospital Fujian Medical University, Fuzhou, Fujian
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of College of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Jinhua People's Hospital, Jinhua, Zhejiang
  - Yuyao People's Hospital, Yuyao, Zhejiang